CLINICAL TRIAL: NCT05145582
Title: Role of Online Discussion Forums in Unguided Internet-Delivered Cognitive Behavioural Therapy for Canadian Public Safety Personnel: A Randomized Trial
Brief Title: Exploring the Role of Online Discussion Forums in Internet-Delivered Therapy for Canadian Public Safety Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Government of Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-130
Record Dates: First submitted 2021-11-17; First posted 2021-12-06 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Depression; Anxiety; Stress Disorders, Post-Traumatic
Keywords: Internet-Based Intervention; Cognitive Behavioral Therapy; Telemedicine
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two treatment conditions (unguided ICBT only or unguided ICBT + online discussion forum)
Masking Description: Participants cannot be blinded to condition because ICBT (like other psychotherapies) cannot be both provided to and concealed from a participant. However, the difference between the two conditions (i.e., presence or absence of an online discussion forum) will be concealed from all participants. Because only participants assigned to the ICBT + Peer Support Forum condition will have access to the Peer Support Forum, it will not be possible to mask the forum moderator to those participants' condition. Because outcomes will be assessed via self-report questionnaire measures, outcomes assessor masking is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unguided, Transdiagnostic ICBT Tailored for PSP (Experimental): An 8-week, unguided, transdiagnostic ICBT program tailored specifically for public safety personnel and designed to treat depression, anxiety, and PTSD.
  Interventions: Behavioral: The Self-Guided PSP Wellbeing Course
- Unguided, Transdiagnostic ICBT Tailored for PSP + Online Discussion Forum (Experimental): An 8-week, unguided, transdiagnostic ICBT program tailored specifically for public safety personnel and designed to treat depression, anxiety, and PTSD plus a built-in online discussion forum.
  Interventions: Behavioral: The Self-Guided PSP Wellbeing Course; Behavioral: Online Discussion Forum

INTERVENTIONS:
Behavioral: The Self-Guided PSP Wellbeing Course — An unguided version of a transdiagnostic ICBT program that has shown promising initial outcomes in prior research (https://doi.org/10.2196/27610).
Behavioral: Online Discussion Forum — An online discussion forum designed to provide an opportunity for participants to support one another in their use of the ICBT program.
  Arms: Unguided, Transdiagnostic ICBT Tailored for PSP + Online Discussion Forum

SUMMARY:
This study is a randomized trial designed to evaluate unguided (i.e., purely self-help), transdiagnostic internet-delivered cognitive behavioural therapy tailored specifically for public safety personnel both with and without a built-in online discussion forum.

DETAILED DESCRIPTION:
--------------

Background:

--------------

The investigators' research unit, PSPNET, is currently providing therapist-guided internet-delivered cognitive behavioural therapy (ICBT) to public safety personnel (PSP) in the Canadian provinces of Saskatchewan, Quebec, Nova Scotia, and New Brunswick. Specifically, PSPNET is offering PSP a transdiagnostic ICBT program for depression, anxiety, and PTSD (the PSP Wellbeing Course), as well as a disorder-specific ICBT program for PTSD (the PSP PTSD Course). ICBT is effective and can help overcome many of the barriers to traditional, face-to-face mental healthcare that PSP face (e.g., concerns about privacy, stigma, distance from services, cost of treatment).

The investigators have created an unguided version of the PSP Wellbeing Course (i.e., no therapist guidance) called the Self-Guided PSP Wellbeing Course. They plan to evaluate this ICBT program through a randomized trial across Canada. Although unguided ICBT does not tend to be quite as effective as guided ICBT, it still consistently results in favorable outcomes compared with control conditions. An important advantage of unguided ICBT is its greater scalability-that is, once created, an unguided ICBT program can be delivered easily on a large scale. Given that PSP face many barriers to mental healthcare, it is expected that participation in this study will help extend treatment to individuals who have not been able to access traditional, face-to-face mental healthcare services. Further, participants will be free to access any other services they see fit while participating in this research.

Prior studies evaluating unguided ICBT interventions that have included online discussion forums have demonstrated excellent results, in many cases finding outcomes comparable to those found in trials of guided ICBT and face-to-face therapy. However, no prior study has experimentally tested the impact of adding an online discussion forum to an unguided ICBT intervention.

The objectives of this new proposed study are (a) to evaluate the first-ever transdiagnostic, unguided ICBT program tailored for PSP, (b) to conduct the first experiment assessing whether a therapist-moderated online discussion forum (hereafter described as the "Peer Support Forum", as it will be known to participants) affects outcomes, and (c) to conduct a mixed-methods analysis of participant feedback on the discussion forum to inform future efforts to implement discussion forums in ICBT. This will be done using a randomized trial comparing the Self-Guided PSP Wellbeing Course with a version of the Self-Guided PSP Wellbeing Course that includes the Peer Support Forum. Participants assigned to the condition with the Peer Support Forum will be encouraged to discuss the course with each other and support one another in using it throughout their participation in the study.

This project is expected to have four implications: (a) to provide treatment to the PSP who participate in it; (b) to inform the potential future use of unguided ICBT for PSP; (c) to experimentally assess whether adding an online discussion forum to an unguided ICBT intervention improves outcomes, and (d) to assess what participants like and dislike about online discussion forums within the context of an ICBT intervention to help guide the future implementation of online discussion forums in ICBT.

--------------

Overview of Methods:

--------------

The proposed research will consist of a randomized trial (N = 114) with two conditions, both of which will involve an eight-week, transdiagnostic unguided ICBT intervention tailored for Canadian PSP. One condition will consist of the ICBT intervention only ("ICBT-Only condition"), and the other will consist of the ICBT intervention with a therapist-moderated online discussion forum ("ICBT + Peer Support Forum condition"). Participants will be administered a battery of self-report measures during eligibility screening and at eight and 20 weeks post-enrollment. Primary outcomes will include changes in symptoms of depression, anxiety, and posttraumatic stress disorder. Secondary outcomes will include treatment satisfaction, treatment engagement, patient-program alliance, and changes in health service use, resilience, subjective wellbeing, and functional impairment. Treatment outcomes will be compared across the two conditions using multilevel modeling. The investigators will also use qualitative analysis to further examine treatment satisfaction and participants' experiences with the Peer Support Forum. Of note, the sample size (N = 114) was calculated as a minimum acceptable sample size, and the investigators plan to recruit more participants if possible, given the uncertainty around the size of effect they may ultimately find.

--------------

Measures:

* Change in symptoms of depression (PHQ-9)
* Change in symptoms of anxiety (GAD-7)
* Change in symptoms of PTSD (PCL-5)
* Change in resilience (BRS)
* Change in wellbeing (FS)
* Change in healthcare use (Healthcare Use Questionnaire)
* Treatment satisfaction (Treatment Satisfaction Questionnaire)
* Patient-program alliance (SRS)
* Demographic information (Participant Information Questionnaire)
* Knowledge and perceptions of ICBT)
* Alcohol use (AUDIT)
* Drug use (DUDIT)

Procedure:

--------------

To enroll in the proposed study, PSP will access a study web page that will provide some basic information about the study. Interested PSP will then click a link to access the study consent form. It is not possible for participants to be blinded to their condition in psychotherapy research, but the consent form will describe the study only in general terms (e.g., it will not mention the Peer Support Forum) so that each participant can be kept blind to how their condition differs from others. Prospective participants who provide informed consent will be administered the Participant Information Questionnaire, PHQ-9, GAD-7, PCL-5, BRS, FS, AUDIT, DUDIT, Health Service Use Questionnaire (screening version), and ICBT Feedback Questionnaire. Prospective participants who are under the age of 18 will immediately and automatically be notified that they are ineligible to participate. Otherwise, participant eligibility will be reviewed by the principal investigator and/or a research assistant. Eligible participants will be randomly assigned to conditions using the website randomizer.org and manually enrolled in one of the two versions of the Self-Guided PSP Wellbeing Course (i.e., the ICBT-Only version or the ICBT + Peer Support Forum version). Due to concerns that psychosis, mania, or substance abuse could interfere with participants' ability to engage in the Peer Support Forum in a constructive way, eligible participants reporting these characteristics will be nonrandomly assigned to the ICBT-Only condition and excluded from the main analyses.

Participants will receive an email informing them that they have been assigned to a condition and may begin the Self-Guided PSP Wellbeing Course on the next Monday. Individuals who are ineligible to participate but 18 years of age or older will receive an email informing them that they are ineligible to participate in the study but may receive access to the treatment content without being part of the study if they wish. This procedure is expected to provide a disincentive for prospective participants who are deemed ineligible to attempt to enroll again using deceptive responses to the screening questionnaires. The investigators will send login information to participants and nonparticipants who are given access to the treatment materials by email. Upon logging in for the first time, prospective participants will immediately be prompted to change their passwords. Participants will be given access to the Self-Guided PSP Wellbeing Course, and participants assigned to the ICBT + Peer Support Forum condition will be given access to it through a link embedded in their version of the course. Before accessing the Peer Support Forum, they will be required to provide informed consent to engage in the Peer Support Forum and agree to the Forum Terms of Use.

Eight weeks after their date of enrolment-and again at 20 weeks after their date of enrolment-participants will receive an automated email asking them to complete posttreatment questionnaires. Participants will provided informed consent to continue their participation in the study before completing these questionnaires. The posttreatment questionnaires will include the PHQ-9, GAD-7, PCL-5, BRS, and FS. At eight weeks, but not at 20 weeks, participants will also be asked to complete the Health Service Use Questionnaire (posttreatment version), adapted SRS, and Treatment Satisfaction Questionnaire. Participants will be asked to complete these measures within four weeks of them being made available. Participants will also be asked to complete an extremely brief Program Usage Questionnaire at 2, 4, 6, and 8 weeks. Participants will be able to access the Self-Guided PSP Wellbeing Course (and the Peer Support Forum, for participants who are granted access to it) for 20 weeks after their date of enrolment.

--------------

Peer Support forum:

--------------

All participants assigned to the ICBT + Peer Support Forum condition will be given access to the same forum (i.e., there will not be multiple forums). The Peer Support Forum will be moderated by the principal investigator, with support from PSPNET's team of registered therapists as necessary. The principal investigator will check the forum daily and post comments as appropriate to facilitate discussion. The number of comments the principal investigator will post and the amount of time spent moderating the Peer Support Forum will depend on the level of activity in the forum and will be documented and reported. The principal investigator has a master's degree in clinical psychology.

The Peer Support Forum will include a Terms of Use page that will be prominently displayed for participants to review. The forum will include several sections, and participants will not be able to add new sections. Within each section, however, participants will be able to add topics and respond to topics via posts. That is, posts are nested within topics, which are in turn nested within sections. The Peer Support Forum will include the following seven sections: one for each of the five lessons of the Self-Guided PSP Wellbeing Course, one for clients who have completed all lessons, and a miscellaneous section. Additional sections may be added during the course of the study as necessary.

In addition to being able to create topics and posts in the Peer Support Forum, participants will be able to flag posts to alert the moderating therapist to inappropriate content. Flagged posts will be hidden until the moderator reviews them, with a note stating that they have been flagged due to a potential violation of the Terms of Use. The moderator will then decide whether a flagged post is in violation of the Terms of Use, in which case it will remain hidden, or whether it should be made visible again. Participants will also be able to create nicknames for themselves that will appear on the topics and posts they create. The Terms of Use urge participants to avoid using any self-identifying information within their chosen nickname. If a participant chooses a nickname that reveals their identity, a member of the PSPNET team will email the participant to ask them to change it.

ELIGIBILITY:
Inclusion Criteria

* At least 18 years of age
* Current or former public safety personnel (or public safety personnel trainee)
* Residing in Canada at time of enrollment
* Has regular access to the internet

Exclusion Criteria

* Not 18 years of age or older
* Not a current or former public safety personnel (or public safety personnel trainee)
* Not residing in Canada at time of enrollment
* Does not have regular access to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Depression | Baseline, 8 weeks, 20 weeks
  Patient Health Questionnaire-9. The Patient Health Questionnaire-9 (PHQ-9) is a commonly used measure of depression that includes an item to measure suicidality (Kroenke et al., 2001). It has demonstrated excellent psychometric properties in many studies (e.g., Cameron et al., 2008; Kroenke et al., 2001, 2010). Its nine items are rated on a four-point Likert scale from 0 (not at all) to 3 (nearly every day) for a total score ranging from 0 to 27. Traditionally, a score of 10 or greater has been considered indicative of a likely diagnosis of major depressive disorder on the PHQ-9 (Manea et al., 2012). A change in score of six points has been identified as a reliable change index (National Collaborating Centre for Mental Health, 2019).
Change in Anxiety | Baseline, 8 weeks, 20 weeks
  Generalized Anxiety Disorder-7. The Generalized Anxiety Disorder-7 (GAD-7) is a seven-item measure of generalized anxiety symptoms. Like the PHQ-9, its items are rated on a four-point Likert scale from 0 (not at all) to 3 (nearly every day). Possible total scores range from 0 to 21. Research shows that the GAD-7 has strong psychometric properties, and a score of 10 or greater can be used to indicate a likely diagnosis of generalized anxiety disorder (Kroenke et al., 2010; Spitzer et al., 2006). Following the precedent of other ICBT researchers, a change in score of five points or more will be considered clinically significant (Titov et al., 2017).
Change in Posttraumatic Stress | Baseline, 8 weeks, 20 weeks
  PTSD Checklist for DSM-5. The PTSD Checklist for DSM-5 (PCL-5) is a common measure of PTSD that was updated following the release of the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5; (American Psychiatric Association, 2013; Blevins et al., 2015; Weathers et al., 2013). It includes 20 items that are rated on a five-point Likert scale from 0 (not at all) to 4 (extremely), for a total score between 0 and 80. Several research groups have suggested that a score of 33 or greater indicates a likely diagnosis of PTSD (Bovin et al., 2016; Wortmann et al., 2016). A change in score of 10 points or more is considered a reliable change on the PCL-5 (Byllesby et al., 2019). At baseline (but not at later timepoints), the investigators will administer a version of the PCL-5 that includes five additional questions about the nature of the potentially psychologically traumatic event that a respondent experienced (Weathers et al., 2013).

SECONDARY OUTCOMES:
Change in Functional Impairment | Baseline, 8 weeks, 20 weeks
  Sheehan Disability Scale. The Sheehan Disability Scale (SDS) is a three-item measure of functional impairment that has demonstrated good psychometric properties (Sheehan, 1983). Each item inquires about the degree to which symptoms have disrupted a different domain in a respondent's life (i.e., work/school, social life, and family life/home responsibilities). Response options range from 1 (not at all) to 10 (extremely) on a visual analog scale. The items can be interpreted individually or summed for a total score between 0 and 30. There is no clinical cut-off score.
  Of note, although we originally planned to administer the SDS, we ultimately removed it from our outcome measures because we were unable obtain permission to use it.
Change in Resilience | Baseline, 8 weeks, 20 weeks
  Brief Resilience Scale. The Brief Resilience Scale (BRS) is a six-item self-report measure of resilience that has demonstrated good reliability and validity (Leontjevas et al., 2014; Smith et al., 2008; Windle et al., 2011). Responses are selected using a five-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), and a higher mean score indicates greater resilience. Three of the items are reverse-scored.
Change in Wellbeing and Flourishing | Baseline, 8 weeks, 20 weeks
  Flourishing Scale. The Flourishing Scale (FS) is an eight-item self-report measure of flourishing across several important domains of human functioning (e.g., positive relationships, meaning and purpose, feelings of competence). The FS has demonstrated good psychometric properties and correlates strongly with other measures of wellbeing (Diener et al., 2009, 2010). Responses are selected using a seven-point Likert scale from 1 (strongly disagree) to 7 (strongly agree) for a total score between 8 and 56. It is worth noting that the FS was formerly called the Psychological Well-Being Scale, but its name was changed to reflect its measurement of a construct broader than wellbeing as it is commonly defined (Diener et al., 2010). A higher score indicates a higher degree of flourishing across various facets of human life.
Change in Healthcare Use | Baseline, 8 weeks, 20 weeks
  Healthcare Use Questionnaires. The Healthcare Use Questionnaires will be administered during eligibility screening, and a different version of this questionnaire will be administered at eight weeks and 20 weeks. Both versions will include a series of questions related to participants' past and current use of healthcare services, particularly for mental health challenges.
Treatment Satisfaction | 8 weeks
  Treatment Satisfaction Questionnaire. The Treatment Satisfaction Questionnaire is a brief bespoke questionnaire assessing participants' treatment satisfaction. Participants assigned to the ICBT + Peer Support Forum condition will be presented with an expanded version of this questionnaire that will include questions assessing their satisfaction and experiences with the forum.
Patient-Program Alliance | 8 weeks
  Adapted Session Rating Scale. The Session Rating Scale (SRS) is a four-item scale originally designed to measure clients' perceptions of the working alliance between themselves and their therapists (Miller et al., 2000). The items assess perceptions of bond, goal agreement, task agreement, and overall working alliance. They are rated on a seven-point Likert scale from 0 (absolutely disagree) to 6 (absolutely agree). The SRS has demonstrated good psychometric properties (Campbell & Hemsley, 2009; Duncan et al., 2003). Cavanagh and colleagues (2018) adapted the SRS to measure patient-program alliance in an ICBT study. The investigators will use their adapted version of the SRS with a slight wording change to each item, such that the measure refers to the Self-Guided PSP Wellbeing Course by name.
Program Use | 2 weeks, 4 weeks, 6 weeks, 8 weeks
  Program Use Questionnaire. This is a two-item bespoke questionnaire assessing the degree to which participants engaged with treatment content and the degree to which they found it helpful during the course of treatment. Participants assigned to the ICBT + Peer Support Forum condition will receive an additional three items assessing the degree to which they engaged with the forum and the degree to which they found it helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh C McCall, MA, Principal Investigator — University of Regina; Heather D Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (2):
- Canada (2):
  - Department of Psychology and Collaborative Centre for Justice and Safety, Regina, Saskatchewan
  - University of Regina, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCall HC, Hadjistavropoulos HD. Impact of an Online Discussion Forum on Self-Guided Internet-Delivered Cognitive Behavioral Therapy for Public Safety Personnel: Randomized Trial. J Med Internet Res. 2024 Aug 14;26:e59699. doi: 10.2196/59699. PMID 39141899